CLINICAL TRIAL: NCT06908902
Title: Prospective Study on the Safety and Efficacy of Robot-Assisted Laparoscopic Partial Nephrectomy With Renal Artery Off-Clamp in the Treatment of cT1 Renal Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-sr-972
Record Dates: First submitted 2024-12-11; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: RCC, Renal Cell Cancer; Partial Nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- renal artery block-off set (Experimental)
  Interventions: Procedure: partial nephrectomy with zero renal artery clamping
- renal artery block set (Active Comparator)
  Interventions: Procedure: partial nephrectomy with main or branch renal artery clamping

INTERVENTIONS:
Procedure: partial nephrectomy with main or branch renal artery clamping — Robotic-assisted laparoscopic or laparoscopic partial nephrectomy with main or branch renal artery clamping
  Arms: renal artery block set
Procedure: partial nephrectomy with zero renal artery clamping — Robotic-assisted laparoscopic partial nephrectomy with zero renal artery clamping
  Arms: renal artery block-off set

SUMMARY:
Renal tumors are common urological cancers, with over 430,000 new cases and more than 170,000 deaths globally in 2020. In China, renal cancer ranks third among urological malignancies, with an increasing incidence. Risk factors include smoking, obesity, hypertension, and family history. Surgery, including partial nephrectomy and radical nephrectomy, is the primary treatment. According to AJCC staging, tumors ≤7 cm confined to the kidney are classified as T1 stage. Studies show no significant difference in cancer-specific survival between partial nephrectomy and radical nephrectomy for T1 tumors, and partial nephrectomy preserves renal function, reducing the risk of metabolic and cardiovascular diseases. Therefore, European guidelines recommend partial nephrectomy for cT1a-b tumors.

Partial nephrectomy can be performed via open surgery, laparoscopy, or robotic assistance, each with pros and cons. Robotic or laparoscopic approaches have less blood loss and shorter hospital stays compared to open surgery. A 7-year follow-up shows no significant difference in oncological outcomes. The surgical goal is to remove the tumor with negative margins while preserving normal renal tissue. Factors such as preoperative renal function, ischemia time, extent of normal tissue resection, blood loss, and suturing technique affect postoperative renal function.

Renal artery clamping is often required during partial nephrectomy to improve visibility, but it leads to ischemia-reperfusion injury, so minimizing damage is crucial. Controlling warm ischemia time is an effective strategy, with guidelines recommending ischemia time under 30 minutes. Studies show that continuous or knotless suturing techniques reduce ischemia time and blood loss. Additionally, minimizing the ischemic area helps protect renal function. Our center explored branch renal artery clamping, which, although increasing ischemia time, better protects kidney function. A study showed a smaller decline in glomerular filtration rate (GFR) with branch clamping compared to conventional clamping.

Gill et al. reported a "zero-ischemia" technique using controlled hypotension and selective clamping of higher-level renal artery branches, showing no significant change in serum creatinine or GFR. However, both renal artery clamping techniques cause ischemia-reperfusion injury, affecting renal function. A study of robotic-assisted partial nephrectomy found that 20.2% of patients had worsened chronic kidney disease (CKD) staging, with statistically significant differences in preoperative and postoperative GFR and CKD staging.

For patients with solitary or functionally solitary kidneys, or those with comorbidities like hypertension or diabetes, renal artery clamping may worsen acute renal dysfunction and increase the risk of long-term kidney failure. Avoiding renal artery clamping may reduce ischemia-reperfusion injury, but its safety and efficacy remain unclear.

A retrospective study of 537 solitary kidney patients undergoing open surgery with different vascular management strategies (no clamping, warm ischemia, and cold ischemia) showed that the risk of renal failure was lower in patients without ischemia. While this study focused on open surgery, it raises the question of whether zero-ischemia partial nephrectomy is feasible in minimally invasive surgery. A study on 141 renal angiomyolipoma patients using a zero-ischemia technique showed no significant change in GFR. However, this method may not be suitable for malignant tumors.

the investigators aims to evaluate whether robotic-assisted laparoscopic partial nephrectomy using a zero-ischemia technique for cT1 renal tumors can better protect renal function, reduce postoperative complications, and not affect oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Imaging examination confirms a T1 renal tumor (including T1a and T1b), and the investigator deems partial nephrectomy to be beneficial.
* Age ranges from 18 to 90 years.
* No history of severe kidney disease or autoimmune disorders.
* Cardiopulmonary function indicates the ability to tolerate major abdominal surgery.
* ECOG performance status score is 0 or 1.
* Willingness to undergo zero-ischemia partial nephrectomy and able to provide written informed consent, understanding and agreeing to comply with the study requirements and evaluation schedule.

Exclusion Criteria:

* Imaging assessment shows a tumor stage of ≥T2.
* Imaging indicates that the tumor is located in the renal pelvis or is a Wilms' tumor, etc.
* The investigator considers the patient unsuitable for partial nephrectomy.
* Major surgery or significant trauma occurred within 28 days prior to enrollment.
* Live vaccine received within 28 days prior to enrollment.
* Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral treatment occurred within 14 days prior to enrollment.
* Any traditional Chinese medicine or herbal supplements for cancer treatment taken within 14 days prior to enrollment.
* Participation in any other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
serum creatinine | Preoperative serum creatinine and Serum creatinine at 3 days postoperative;

SECONDARY OUTCOMES:
Recurrence-Free Survival（RFS） | From enrollment to 3 years post-treatment completion
Glomerular Filtration Rate（GFR） | GFR before the surgery and GFR at 1 month, 3 months, and 12 months postoperative.

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China